CLINICAL TRIAL: NCT07010627
Title: Evaluation of the Application of Auricular Laserpuncture in the Treatment of Chronic Pain
Brief Title: Chronic Pain Treatment Whith Auricular Laserpuncture
Status: Enrolling by invitation | Type: Observational
Sponsor: Universidade do Vale do Paraíba (Other)
Collaborators: Ministry of Education, Brazil (Other Government)
Responsible Party: Sponsor
Other Study IDs: 78513124.1.0000.5503
Record Dates: First submitted 2025-04-23; First posted 2025-06-08 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Chronic Knee Pain; Chronic Shoulder Pain; Chronic Low Back Pain
Keywords: chronic pain; elderly; auricular laserpuncture; auriculotherapy
MeSH Terms: conditions — Chronic Pain | interventions — Auriculotherapy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Auriculotherapy for chronic pain treatment with laser stimulation of acupoints using red light: "Stimulation using a laser programmed in continuous mode, emitting red light (4 J of energy) at the following auricular acupoints:
  1. Chronic shoulder pain: shen men, kidneys, peripheral nervous system, analgesia, muscle relaxation, shoulder region, adrenal;
  2. Chronic knee pain: shen men, kidneys, peripheral nervous system, analgesia, muscle relaxation, knee region, adrenal;
  3. Chronic lumbar pain: shen men, kidneys, peripheral nervous system, analgesia, muscle relaxation, lumbar region, adrenal."
  Interventions: Procedure: Auriculotherapy for chronic pain treatment with laser stimulation of acupoints using red light
- "Auriculotherapy for chronic pain treatment with stimulation of acupoints using mustard seeds.": The conventional clinical practice treatment will be carried out, consisting of the application of mustard seeds to stimulate the following auricular acupoints:
  1. Chronic shoulder pain: shen men, kidneys, peripheral nervous system, analgesia, muscle relaxation, shoulder region, adrenal;
  2. Chronic knee pain: shen men, kidneys, peripheral nervous system, analgesia, muscle relaxation, knee region, adrenal;
  3. Chronic lumbar pain: shen men, kidneys, peripheral nervous system, analgesia, muscle relaxation, lumbar region, adrenal.
  Interventions: Procedure: "Auriculotherapy for chronic pain treatment with stimulation of acupoints using mustard seeds."

INTERVENTIONS:
Procedure: Auriculotherapy for chronic pain treatment with laser stimulation of acupoints using red light — This arm of the study will analyze the effectiveness of the treatment protocol for chronic pain in the shoulder, knee, or lumbar spine region in elderly individuals, using the application of laser acupuncture with low-power laser and red light on acupoints of Auriculotherapy.
  As a criterion for the qualitative evaluation of the study, the McGill questionnaires (Annex A) and the Visual Analog Scale (Annex B) will be used to assess chronic pain, while the SF-36 instrument (Annex C) will allow for the evaluation of participants' quality of life before and after the treatment protocol.
  For quantitative evaluation, thermographic images and the Ryodoraku System will be used. All proposed tools will be applied before the first treatment session (A1), before the fifth session (A2), and at the end of the tenth session (A3).
  Groups: Auriculotherapy for chronic pain treatment with laser stimulation of acupoints using red light
Procedure: "Auriculotherapy for chronic pain treatment with stimulation of acupoints using mustard seeds." — This arm of the study will analyze the effectiveness of the treatment protocol for chronic pain in the shoulder, knee, or lumbar spine regions in elderly individuals, utilizing the application of mustard seeds on Auriculotherapy acupoints.
  As criteria for the qualitative evaluation of the study, the McGill questionnaires (Annex A) and the Visual Analog Scale (Annex B) will be used to assess chronic pain, while the SF-36 instrument (Annex C) will allow for the evaluation of participants' quality of life before and after the treatment protocol.
  For quantitative evaluation, thermographic images and the Ryodoraku System will be utilized. All proposed tools will be applied before the first treatment session (A1), before the fifth session (A2), and at the end of the tenth session (A3)
  Groups: "Auriculotherapy for chronic pain treatment with stimulation of acupoints using mustard seeds."

SUMMARY:
The objective of the study to evaluate the effectiveness of a treatment protocol using auricular acupuncture point stimulation with laser , compared to the use of mustard seeds, for reducing chronic pain in the elderly. With this research, the researches hope to obtain results that allow us to establish a non-invasive, easy, quick-to-apply, and painless treatment protocol to minimize chronic pain in the lumbar spine, shoulders, and knees, thereby improving the quality of life of the target population in this study.

In the first session and before the start of the treatment protocol, three questionnaires will be applied for evaluation of the subjects: the first to assess quality of life (SF-36), and the others to evaluate pain intensity (Visual Analog Scale for pain and the McGill Pain Questionnaire). The pain location will be assessed using a thermografic camara that evaluates skin temperature, as well as a Traditional Chinese Medicine device (Ryodoraku) that measures the energy flow in the body's meridians. The same evaluation protocol will be repeated before the fifth session and after the tenth session.

DETAILED DESCRIPTION:
This study will analyze the effectiveness of treatment protocols A or B for chronic pain in the shoulder, knee, or lumbar spine regions in elderly individuals. The protocol A involves the application of low-power red laser therapy on auriculotherapy acupoints. The protocol B involves the application of mustard seeds . To assess the qualitative aspect of the study, the McGill Pain Questionnaire and the Visual Analog Scale will be used to evaluate chronic pain, while the SF-36 instrument will assess the participants' quality of life before and after the treatment protocol. For the quantitative evaluation, thermographic imaging and the Ryodoraku System will be used. All proposed tools will be applied before the first treatment session, before the fifth session ,and at the end of the tenth session.

Risks and Benefits During the study, participants will be subject to risks related to physical and psychological discomfort due to the proposed therapeutic protocol. All procedures will be performed individually in an appropriate and private room to ensure the participant's comfort and privacy. Each participant will be provided with protective goggles, which must be worn throughout the laser application period. These goggles will be sanitized before each session, and the laser device tip will be covered with PVC film, replaced after each session.

Although rare, stimulation of the auricular pavilion may cause transient side effects such as local pain, fatigue, dizziness, nausea, and headaches. The use of the laser may generate slight discomfort, such as mild warming, but this effect is temporary and has no serious consequences. If a participant experiences any of these symptoms or any other physical discomfort, the protocol will be immediately interrupted, and the participant will remain under observation by the researcher until they feel better. The use of mustard seeds may cause mild pain at the application site, but this typically subsides over time. Participants will be informed that if a seed falls off prematurely, it will not affect the treatment, and they should continue stimulating the remaining seeds three times a day and remove them one day before the next session.

Psychological discomfort may also arise when participants answer the questionnaires. The questionnaire will be administered in a private setting with only the participant and the researcher present. If the participant feels uncomfortable, they may request to withdraw from the study.

To minimize the risk of exposure of participants' personal data, the researcher commits to storing all collected data in password-protected digital files accessible only to the research team. Each participant will be assigned an individual identification code to prevent any possibility of access or identification.

Whenever the participant wishes, the principal researcher will provide clarifications regarding the procedures to establish trust. Participants will be informed that they may withdraw from the study at any time without affecting the continuity of their treatment.

As a benefit of this study, the results are expected to help establish a non-invasive, easy-to-apply, and ergonomically comfortable treatment protocol for chronic pain in elderly individuals, thereby improving their quality of life.

Clinical Protocol The participant will be received in a private room with only the researcher present. They will be instructed to sit in a chair comfortably. The McGill Pain Questionnaire, the SF-36 questionnaire, and the Visual Analog Scale for Pain will then be administered to assess the intensity of pain and its impact on the participant's quality of life.

After completing the questionnaires, while still seated, the researcher will evaluate the participant using the Ryodoraku System for bioenergetic meridian measurement. This assessment will be conducted through 24 reactive points, known as electro-permeable skin points , located on the upper and lower limbs at the acupoints P9, PC7, C7, ID5, TA4, IG5, BP3, F3, R4, B65, VB40, and E42. The Ryodoraku System is a portable electronic device equipped with two wand-shaped electrodes. One wand will be held by the participant, while the researcher manipulates the other, placing it in direct contact with the acupoints. The device is connected via USB to a computer with pre-installed software, generating graphs that compare the participants' meridian conditions and possible energy imbalances with a standard balanced energy pattern.

Next, thermographic images of the area where the participant experiences chronic pain will be taken using a thermal imaging camera. During this process, participants will stand upright on an insulated rubber surface. The analyzed region must be free of clothing. Images will be captured from a distance of 100 cm from the target area to ensure proper framing, against a black background to avoid infrared radiation reflection. Participants will be instructed to avoid alcohol, physical exercise, bathing, and stimulant intake (such as caffeine) for at least two hours before the examination.

The evaluation tools for research data collection will be applied before the first session , before the fifth session , and after the tenth session .

Treatment Protocol For participants in Group A (GA), a portable Recover laser device (MMO, with LI-Ion 7.4V/650 mA battery, ) will be used. This device emits visible and invisible laser radiation, with a diode laser λ=600 nm/808 nm, P=100mW (each laser), , programmed in continuous mode with red light emission at 4 J power. All participants will sit in a comfortable position and wear protective goggles provided by the researcher (who will also wear goggles during laser application).

For participants in Group B , mustard seeds will be applied with micropore tape to the same auriculotherapy acupoints used in group A. Each participant will undergo ten sessions, twice a week, over five weeks of treatment.

The auriculotherapy acupoints will be located in the right auricular pavilion for all participants. These points will be previously cleaned with gauze soaked in 70% alcohol. Additionally, the laser device tip will be wrapped in PVC film, which will be replaced for each participant.

ELIGIBILITY:
Inclusion Criteria

* Participants aged between 60 and 90 years;
* Both sexes;
* Report of chronic pain in the lumbar region, shoulders, or knees;
* Sign the Informed Consent Form.

Exclusion Criteria:

* Undergoing treatment similar to the proposed research protocol at another facility or physiotherapy service;
* Using analgesic or anti-inflammatory medications;
* Unable to fully understand the protocol proposed by the researcher;
* Unwilling to participate in the study and/or unavailable to attend all proposed treatment sessions;
* Presence of lesions on the auricular pavilion;
* Wearing earrings or piercings in the acupoint regions targeted for laser stimulation.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Initially, in order to recruit participants for this study, invitation flyers will be displayed at the Castejon Campus, home to the Faculty of the Third Age, and at the Urbanova Campus, home to the Faculty of Health Sciences (FCS), both part of the University of Vale do Paraíba (UNIVAP), located in São José dos Campos, Brazil.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Comparative efficacy evaluation between the application of auricular laser acupuncture and the use of mustard seeds in the treatment of chronic pain | Untill the completion of the study which take approximately 12 months
  The collected data will be entered and tabulated in Excel 2010 and analyzed using the Statistical Package for the Social Sciences (SPSS), version 17.0. The Shapiro-Wilk test will be performed on numerical variables to determine whether they follow a normal distribution. A significance level of 0.05 will be adopted to assess normality. For normally distributed data, Pearson's correlation coefficient (r) will be used to measure the magnitude and degree of relationship between variables, and Student's t-test will be applied to evaluate significant differences between the means of two conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Luís Eduardo S soares, co-advisor doctoral, Study Director — UNIVAP- University of Paraiba Valley; Emilia Angela A arisawa, advisor doctoral, Study Director — UNIVAP- University of Paraiba Valley; Gerson Q Quadros Jr, Doctoral Student, Principal Investigator — UNIVAP- University of Paraiba Valley
Locations (1):
- UNIVAP- University of Paraiba Valley, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Description of the IPD to be Shared:
  All individual participant data (IPD) collected during the study, including de-identified demographic data, clinical outcomes (pain scores, quality of life assessments), Ryodoraku measurements, and thermographic imaging data.
  What data will be shared:
  All IPD underlying the results of the published primary and secondary outcome measures.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: When will the data be available:
  6 months after the publication of the main results.
  How long will the data be available:
  The data will be available for 5 years after the initial publication.
Access Criteria: Qualified researchers who submit a methodologically sound proposal for secondary analyses.